CLINICAL TRIAL: NCT02942680
Title: A Prospective Randomized Study of the Efficacy and Safety of Aspirin Therapy With CABG
Brief Title: Efficacy and Safety of Aspirin Therapy With CABG
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1184
Record Dates: First submitted 2016-01-31; First posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-06

CONDITIONS: Coronary Heart Disease
Keywords: coronary artery bypass grafting
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): acetylsalicylic acid started for 24 hours before surgery and determination of platelet function
  Interventions: Drug: acetylsalicylic acid started for 24 hours before surgery
- Control (Other): acetylsalicylic acid stayed for 5 days before surgery and determination of platelet function
  Interventions: Drug: acetylsalicylic acid stayed for 5 days before surgery

INTERVENTIONS:
Drug: acetylsalicylic acid started for 24 hours before surgery
  Arms: Experimental
Drug: acetylsalicylic acid stayed for 5 days before surgery
  Arms: Control

SUMMARY:
evaluate the safety of preoperative aspirin therapy when performing bypass surgery in conditions of artificial blood circulation

DETAILED DESCRIPTION:
The hypothesis of the study was that aspirin therapy started 24 hours before CABG is safe.

The effectiveness of this hypothesis will be assessed by the presence of a 30-day period after CABG myocardial infarction, ischemic stroke, repeat revascularizations

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Patient able to give informed consent

Exclusion Criteria:

* Missing consent
* Urgent or emergent surgery
* Off-pump CABG
* Рatient has clear indication for anticoagulation (eg. mechanical heart valve, atrial fibrillation) or ADP receptor antagonist (eg. drug-eluting stent)
* History of bleeding diathesis, significant GI bleed, ICH, or liver failure
* Allergy to or intolerance of aspirin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
on discharge drains after surgery in milliliters | 24 hours after surgery

SECONDARY OUTCOMES:
myocardial infarction | myocardial infarction by 30th day after procedure
ischemic stroke | stroke by 30th day after procedure
repeat revascularization | repeat revascularization within 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alexander M. Chernyavskiy, MD PhD, Study Chair — Academician Ye. Meshalkin Novosibirsk Research Institute of Circulation Pathology Ministry of Health care of Russian Federation
Locations (1):
- Meshalkin State Research Institute of Circulation Pathology, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No